CLINICAL TRIAL: NCT04290182
Title: An Open Phase I/II Study in Patients With Dysphonia and Vocal Fold Scarring to Evaluate Safety, Tolerability and Vocal Function After Surgery With Local Administration of Autologous Mesenchymal Stromal Cells
Brief Title: A Study of Local Administration of Autologous Mesenchymal Stromal Cells in Dysphonic Patients With Vocal Fold Scarring
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Swedish Foundation for Strategic Research (Other)
Responsible Party: Principal Investigator, Stellan Hertegård, Adjunct Professor. MD PhD, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-06160 and 5.1-2019-92069
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-03

CONDITIONS: Hoarseness; Dysphonia; Aphonia; Vocal Fold Scar
Keywords: Vocal fold scar; MSC; dysphonia
MeSH Terms: conditions — Hoarseness; Dysphonia; Aphonia

STUDY DESIGN:
Intervention Model Description: This is a phase I/IIa open, single-arm clinical study evaluating the safety and tolerability as well as the influence on VF function, of local injection of the autologous MSC product KI-MSC-PL-204, in patients suffering from chronic VF dysfunction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm: MSC administration to vocal fold scar (Experimental): 1 single arm: Local injection of autologus MSC product (KI-MSC-PL-204) into scarred vocal fold (0,5-1 million cellls/Vocal fold, maximum 2 million cells if bilateral vocal fold scar)
  Interventions: Biological: MSC-KI-PL-204

INTERVENTIONS:
Biological: MSC-KI-PL-204 — Autologous MSC product

SUMMARY:
The overall aim of the project is to develop a new method for treatment of untreatable severe hoarseness due to vocal fold scarring by local injection of autologous mesenchymal stromal cells (MSC). At present there is no lasting effective treatment for this condition which results in personal suffering, and often extended sick leave, change of work or unemployement for the patients.

Based on the previous results the investigators expect the autologous MSC product KI-MSC-PL-204 to be a new effective treatment without side effects for many patients with severe hoarseness or aphonia due to vocal fold scarring.

DETAILED DESCRIPTION:
The general aim of the project is to develop a treatment for severe hoarseness due to vocal fold (VF) scarring. Vocal fold scarring can be caused by tumor surgery, radiotherapy, severe inflammation or is early acquired (sulcus vocalis with scar) and results in stiff vocal folds with decreased vibratory capacity and severe deterioration or total loss of voice (aphonia). There is no lasting effective treatment. Bone marrow derived mesenchymal stem cells (MSC) are immunomodulatory, decrease inflammation and improve endogenous healing. After receiving ethical permission the investigators have since 2012 treated 16 patients with manifest vocal fold scarring and severe hoarseness by scar resection and local injection of autologous bone marrow MSC to restore speech. This project was the first in the world to study the effects of MSC treatment of vocal fold scarring in humans. Analysis was made before and up to 12 months post operatively with voice recordings, examination with high speed camera and elasticity measurements of the vocal folds with novel technology. No side effects were found for any patient and for two thirds of the patients with 12 months follow-up the vocal fold function improved and no patient deteriorated.

While cell therapy with autologous MSC was classified according to the Tissue Legislation before 2015, it is now regarded as drug treatment. In accordance with this legislation, the MSC production is now full scale GMP. The investigators have recently received permissions from Swedish Medical Product Agency (DNr 5.1-2019-92069) and from the Regional ethic committee (Drn 2019-06160) for an open Phase I/Il study in patients with severe dysphonia and vocal fold scarring to evaluate safety, tolerability and vocal function after surgery with local administration of autologous mesenchymal stromal cell product KI-MSC-PL-204 as an extended study on 15 patients.

MSC may in the future be used to treat patients with severe hoarseness due to scarring, as well as other damages in the airways.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-65 years with VF scarring and severe voice problems, such as permanent severe hoarseness, complete aphonia or severe voice strain during speech (>1 year) where other treatments have proven ineffective and no alternative treatment is possible.
* No alternative treatment ongoing or planned (phonosurgery with augmentation implantation, voice therapy or other medical treatment).

Exclusion Criteria:

* Active treatment of laryngeal disorder, inflammatory condition of the larynx, or laryngeal/VF papilloma.
* Diagnosed or suspicion of local malignancy or other malignancies, Disease-free period of >5 years after malignant disease (>10 years for local laryngeal cancer).
* Smokers.
* Large scar defects.
* Pregnant or nursing (lactating) women.
* Serological evidence of infection with HIV, HBV, HCV, HTLV and/or syphilis.
* Active ongoing local or systemic infections.
* Ongoing immune suppressive treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of treatment | 3 year
  Number of serious adverse events/ adverse events treatment and conseques

SECONDARY OUTCOMES:
Assessment of VF function by high speed laryngeal/stroboscopy recordings | from baseline to 1 year after treatment.
  Description: Assessment of VF function change from baseline to 1 year after treatment, as evaluated by an expert panel of high speed laryngeal/stroboscopy recordings. (Expert panel catagories: (Improved, unchanged, deteriorated)
Assessment of subjective VHI change (points) | changes from baseline to 1 year after treatement
  Assessment of patient´s subjective VHI (voice handicap index) ratings change (points)
Assessment of Phonation Threshold Pressure changes (cmH2O) | changes from baseline to 1 year after treatment
  Measurements of phonation threshold pressure (PTP) changes from baseline to 1 year after treatment
Assessment of perceptual voice analysis changes (points) | changes from baseline to 1 year after treatment
  Evaluation by an expert panel of perceptual voice parameters, changes from baseline to 1 year after treatment
Assessment of subjective VFI change (points) | from baseline to 1 year after treatment
  Assessment of Vocal fatigue index (VFI) changes from baseline to 1 year after treatment
Assessment of maximum phonation time change (seconds) | from baseline to 1 year after treatment
  Measurements of maximum phonation time change from baseline to 1 year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Patric Scicluna, Clin Research Manager, Study Chair — Karolinska Trial Alliance
Locations (1):
- Karolinska Trial Alliance, Stockholm, Stockholm County, Sweden